CLINICAL TRIAL: NCT05584930
Title: Evaluation of Serum Clusterin and Serum PTX3 Assay During Febrile Aplasia in Children Treated in Pediatric Oncology
Brief Title: Clusterin, Ptx3 and Pediatric Febrile Neutropenia (CluPPFeN)
Acronym: CluPPFeN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-A01750-43
Record Dates: First submitted 2022-10-10; First posted 2022-10-18 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Cancer Childhood; Febrile Neutropenia
MeSH Terms: conditions — Neoplasms; Febrile Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cancer patient (Other): Collection of blood sample
  Interventions: Other: Collection of blood sample

INTERVENTIONS:
Other: Collection of blood sample — * Visit 1 : At inclusion (day 1 of chemotherapy treatment)
  * Visit 2 : Onset of aplasia
  * Visit 3a : day 1 of the 1st febrile aplasia
  * Visit 3b : day 3 of the 1st febrile episode
  * Visit 3c : day 8 of the 1st febrile episode
  * Visit 4a : second febrile episode (after 7 days)
  * Visit 4b : day 3 of the second febrile episode (after 7 days)

SUMMARY:
Febrile aplasia is a common occurrence in children/adults treated with chemotherapy for malignant blood diseases or solid cancers.

This acquired deficiency of immunity mainly causes susceptibility to bacterial and fungal infections, pathogens normally recognized by specific receptors of innate immunity (Pattern Recognition Receptor, PRR).

Thus, the febrile episodes in the context of post-chemotherapy neutropenia can be bacterial or fungal etiology, but can also frequently be related to viral infections, toxic phenomena or other etiologies. In the absence of a discriminating marker, treatment for all these children is based on early, broad-spectrum antibiotic therapy in hospital. Septic shock or even death by refractory septic shock remain, even if they are rare, real complications in pediatric oncology, requiring discriminatory markers for effective management, While trying to reduce the number and duration of hospitalizations for children at low risk for severe febrile aplasia.

It is therefore necessary to identify other markers allowing the earliest possible classification of episodes of febrile aplasia.

A previous study, conducted by our team, PTX3 and febrile aplasia, studied pentraxin 3 (PTX3), a soluble PRR of the pentraxin family that plays a key role in immune surveillance against pathogens. Preliminary results obtained from samples from a cohort of patients treated in adult hematology and pediatric onco-hematology support a prognostic character of PTX3 in the severity of aplasia, with higher elevations of serum protein during episodes of severe sepsis or septic shock (ongoing analyses and interpretations for the adult population). The available data to date on the pediatric cohort are insufficient to conclude on the value of using PTX3. The investigators therefore wish to create a new paediatric cohort, in order to evaluate the PTX3 levels for the paediatric population and also to perform the assay of a new marker, clusterin.

Clusterin (CLU) is an extracellular chaperone protein of constitutive expression. The Innate Immunity team of the National Institute of Health and Medical Research (INSERM) "1307-Scientific Research National Center (CNRS) 6075" unit has shown that Clu binds to extracellular histones and inhibits their inflammatory, thrombotic and cytotoxic properties. The investigators also observed (i) that in adults without severe sepsis neutropenics, low serum levels of Clu at intake and lack of normalization of rates are associated with higher mortality and (ii) Clu levels are inversely correlated with circulating histone levels. All these data suggest that Clu would have a protective role for histone-induced lesions during sepsis independently of antibiotic treatment, opening an innovative therapeutic pathway in the management of severe sepsis.

CluPPFeN is based on the hypothesis that, in a pediatric population with episodes of febrile aplasia, serum Clu and serum PTX3 levels would discriminate between febrile episodes caused by bacterial infection and other etiologies and, As a result, would reduce the consumption of antibiotics, which provide resistance, and the length of hospitalization.

DETAILED DESCRIPTION:
-Primary objective :

Evaluate serum levels CLU levels during febrile neutropenia in children followed for cancer.

-Secondary objective :

1. Evaluate serum levels of CLU at the beginning of non-febrile aplasia and during a possible 2nd febrile peak
2. Evaluate serum PTX3 levels during febrile neutropenia in children followed for cancer
3. Explore the association between CLU, PTX3 and the severity of the aplasia episode
4. Evaluate the association between CLU and PTX3 levels and the type of pathogen found during febrile aplasia
5. Exploration of the diagnostic contribution of CLU and PTX3 in relation to other known parameters of inflammation (including C reactive protein (CRP), procalcitonin (PCT), fibrinogen, interleukin 1 (IL-1), IL-6, IL-10, Tumor Necrosis Factor (TNF-α), CXCL8, IL17)
6. Exploration of genetic polymorphisms predisposing to bacterial and fungal infections (including PTX3 and CLU gene polymorphisms) in the context of febrile aplasia

ELIGIBILITY:
Inclusion Criteria:

* Child under 18 years
* Hospitalized for chemotherapy leading to febrile aplasia
* Signature of the informed consent of the parents or holder of parental authority and consent of the patient

Exclusion Criteria:

* Expected non aplasing chemotherapy
* Child with less than 5 kg body weight at inclusion

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Evaluate serum CLU levels during febrile neutropenia in children followed for cancer | At inclusion
  Serum CLU levels will be estimated at day 1, day 3 and day 8 of febrile aplasia (PNN < 500/mm3). These assessments will also be performed at day 1 of the aplasing chemotherapy course (prior to chemotherapy administration, this value will be considered the reference value). The unit of analysis will be the number of CLU samples included in each scheduled visit.
Evaluate serum CLU levels during febrile neutropenia in children followed for cancer | up to 2 months
  Serum CLU levels will be estimated at day 1, day 3 and day 8 of febrile aplasia (PNN < 500/mm3). These assessments will also be performed at day 1 of the aplasing chemotherapy course (prior to chemotherapy administration, this value will be considered the reference value). The unit of analysis will be the number of CLU samples included in each scheduled visit.

SECONDARY OUTCOMES:
Evaluate serum levels of CLU at the beginning of non-febrile aplasia and during a possible 2nd febrile peak. | up to 2 months
  An estimate of CLU levels at the beginning of non-febrile aplasia (PNN < 500/mm3) as well as after a second episode of fever (2nd febrile peak) beyond day 7 will be made. An estimate of serum CLU levels will also be made at day 3 of the 2nd febrile peak
Evaluate serum PTX3 levels during febrile neutropenia in children followed for cancer | up to 2 months
  Serum levels of PTX3 will be evaluated using the same pattern and assessment methods previously described for CLU.

CONTACTS AND LOCATIONS:
Overall Officials: Coralie MALLEBRANCHE, Dr, Principal Investigator — UH Angers
Locations (1):
- University Hospital of Angers, Angers, France